CLINICAL TRIAL: NCT02418754
Title: A Phase 2, Double-Masked, Randomized, Controlled, Multiple-Dose, Regimen-Ranging Study of the Efficacy and Safety of Intravitreal REGN2176-3 in Patients With Neovascular Age-Related Macular Degeneration
Brief Title: Study of Intravitreal REGN2176-3 in Participants With Neovascular ("Wet") Age-Related Macular Degeneration (AMD)
Acronym: CAPELLA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: No additional efficacy seen with REGN2176-3 over aflibercept alone
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R2176-3-AMD-1417; NCT02603484 (obsolete NCT alias)
Record Dates: First submitted 2015-04-13; First posted 2015-04-16 (Estimated); Results first posted 2020-10-26 (Actual); Last update posted 2020-10-26 (Actual); Status verified 2020-10

CONDITIONS: Neovascular Age-Related Macular Degeneration
MeSH Terms: interventions — aflibercept

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- REGN2176-3 (1 mg: 2 mg) (Experimental): Intravitreal injection of REGN2176-3 (REGN2176 1 mg and REGN3 2 mg) every 4 weeks for 12 weeks. After Week 12, dosing was monthly up to Week 28, then criteria based re-dosing from Week 28-52.
  Interventions: Drug: REGN2176-3
- REGN2176-3 (3 mg: 2 mg) (Experimental): Intravitreal injection of REGN2176-3 (REGN2176 3 mg and REGN3 2 mg) every 4 weeks for 12 weeks. After Week 12, dosing was monthly up to Week 28, then criteria based re-dosing from Week 28-52.
  Interventions: Drug: REGN2176-3
- Intravitreal Aflibercept Injection (IAI) 2 mg (Experimental): IAI every 4 weeks for 12 weeks. After Week 12, dosing was monthly up to Week 28, then criteria based re-dosing from Week 28-52.
  Interventions: Drug: Intravitreal Aflibercept Injection (IAI)
- REGN2176-3 (3 mg: 2 mg) to IAI 2 mg (Experimental): Intravitreal injection of REGN2176-3 (REGN2176 3 mg and REGN3 2 mg) every 4 weeks for 12 weeks. After Week 12, dosing was monthly with IAI 2 mg up to Week 28, then criteria based re-dosing from Week 28-52.
  Interventions: Drug: Intravitreal Aflibercept Injection (IAI)
- IAI 2 mg to REGN2176-3 (3 mg:2 mg) (Experimental): IAI every 4 weeks for 12 weeks. After Week 12, dosing was monthly with REGN2176-3 (REGN2176 3 mg and REGN3 2 mg) up to Week 28, then criteria based re-dosing from Week 28-52.
  Interventions: Drug: REGN2176-3

INTERVENTIONS:
Drug: REGN2176-3
  Arms: IAI 2 mg to REGN2176-3 (3 mg:2 mg); REGN2176-3 (1 mg: 2 mg); REGN2176-3 (3 mg: 2 mg)
Drug: Intravitreal Aflibercept Injection (IAI)
  Other Names: Eylea®
  Arms: Intravitreal Aflibercept Injection (IAI) 2 mg; REGN2176-3 (3 mg: 2 mg) to IAI 2 mg

SUMMARY:
The primary objective of the study was to explore the effect of REGN2176-3 on the Early Treatment Diabetic Retinopathy Scale (ETDRS) best-corrected visual acuity (BCVA) in participants with neovascular age-related macular degeneration (AMD), compared to intravitreal aflibercept injection (IAI) monotherapy.

The secondary objectives of the study were the following:

* To explore the effect of 2 dose levels of IVT REGN2176-3 on anatomical changes of CNV in participants with nAMD compared to IAI monotherapy (at week 12)
* To evaluate if short-term treatment with REGN2176-3 followed by IAI monotherapy offered the same or additional benefit compared to continuous treatment with REGN2176-3. Also to determine if there was benefit in initiating IAI treatment prior to REGN2176-3 compared to continuous treatment with IAI.
* To assess the safety and tolerability of IVT REGN2176-3 in participants with nAMD

ELIGIBILITY:
Key Inclusion Criteria:

1. Men or women ≥50 years of age
2. Active subfoveal CNV secondary to AMD as evidenced by FA in the study eye, as determined by the reading center, including juxtafoveal lesions that affect the fovea
3. BCVA ETDRS letter score of 73 to 24 (20/40 to 20/320) in the study eye at the screening visit
4. Provide signed informed consent

Key Exclusion Criteria:

1. Any prior treatment with anti-VEGF treatment in the study eye
2. Any prior treatment (ie, systemic or ocular treatment) with PDGF or PDGFR inhibitors
3. Dense fibrotic scar or atrophy in the study eye involving the center of the fovea
4. Presence of retinal pigment epithelial tears or rips involving the macula in the study eye
5. Prior vitrectomy in the study eye
6. Any history of macular hole of stage 2 and above in the study eye
7. Any intraocular or periocular surgery within 3 months of day 1 in the study eye, except lid surgery
8. History of corneal transplant in the study eye
9. Evidence of diabetic retinopathy or diabetic macular edema in either eye
10. Positive serum human chorionic gonadotropin/urine pregnancy test at the screening or baseline visit

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 505 (Actual)
Dates: Start 2015-05-05 (Actual); Primary Completion 2016-08-17 (Actual); Study Completion 2017-04-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (84):
- United States (75):
  - Phoenix, Arizona
  - Tucson, Arizona
  - Arcadia, California
  - Beverly Hills, California
  - Irvine, California
  - Mountain View, California
  - Oceanside, California
  - Sacramento, California
  - Santa Ana, California
  - Colorado Springs, Colorado
  - Fort Lauderdale, Florida
  - Fort Myers, Florida
  - Jacksonville, Florida
  - Melbourne, Florida
  - Miami, Florida
  - Plantation, Florida
  - Tampa, Florida
  - Winter Haven, Florida
  - Augusta, Georgia
  - Marietta, Georgia
  - Chicago, Illinois
  - Oak Forest, Illinois
  - Springfield, Illinois
  - Urbana, Illinois
  - Iowa City, Iowa
  - Shawnee Mission, Kansas
  - Lexington, Kentucky
  - Paducah, Kentucky
  - Baltimore, Maryland
  - Towson, Maryland
  - Boston, Massachusetts
  - Jackson, Michigan
  - Southfield, Michigan
  - Minneapolis, Minnesota
  - Florissant, Missouri
  - Lincoln, Nebraska
  - Omaha, Nebraska
  - Las Vegas, Nevada
  - Bloomfield, New Jersey
  - New Brunswick, New Jersey
  - Albuquerque, New Mexico
  - Albany, New York
  - East Setauket, New York
  - Great Neck, New York
  - New York, New York
  - Orchard Park, New York
  - Rochester, New York
  - Asheville, North Carolina
  - Charlotte, North Carolina
  - Cincinnati, Ohio
  - Oklahoma City, Oklahoma
  - Portland, Oregon
  - Kingston, Pennsylvania
  - Monroeville, Pennsylvania
  - Philadelphia, Pennsylvania
  - Florence, South Carolina
  - Ladson, South Carolina
  - West Columbia, South Carolina
  - Rapid City, South Dakota
  - Knoxville, Tennessee
  - Memphis, Tennessee
  - Nashville, Tennessee
  - Abilene, Texas
  - Austin, Texas
  - Dallas, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - McAllen, Texas
  - San Antonio, Texas
  - The Woodlands, Texas
  - Willow Park, Texas
  - Salt Lake City, Utah
  - Burlington, Vermont
  - Fairfax, Virginia
  - Bellevue, Washington
- Japan (9):
  - Akita
  - Asahikawa
  - Chiyoda-ku
  - Fukushima
  - Kawasaki
  - Matsumoto
  - Nagasaki
  - Nagoya
  - Osaka

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 82 sites in US and 11 sites in Japan. A total of 804 participants were screened. Out of 804 participants, 505 were randomized and treated.
Pre-assignment Details: Participants were initially randomized in a 1:2:2 ratio to receive REGN2176-3 (1 mg:2 mg) (REGN2176 1 mg:REGN3 2 mg) or REGN2176-3 (3 mg:2 mg) (REGN2176 3 mg:REGN3 2 mg) or 2 mg intravitreal aflibercept injection (IAI). One eye was under study (the fellow eye was assessed for safety only).
Units Other Than Participants: Study Eyes
Groups:
- Group 1: REGN2176-3 (1 mg:2 mg): Intravitreal injection of REGN2176-3 (REGN2176 1 mg and REGN3 2 mg) every 4 weeks for 12 weeks. At Week 12, Group 1 continued without a secondary randomization. After Week 12, dosing in Group 1 was monthly up to Week 28, then criteria based re-dosing from Week 28-52.
- Group 2: REGN2176-3 (3 mg:2 mg): Intravitreal injection of REGN2176-3 (REGN2176 3 mg and REGN3 2 mg) every 4 weeks for 12 weeks. At Week 12, a secondary randomization occurred in Group 2 for those participants who completed the Week 12 assessments. After Week 12, dosing in Group 2 was monthly up to Week 28, then criteria based re-dosing from Week 28-52.
- Group 3: Intravitreal Aflibercept Injection (IAI) 2 mg: IAI every 4 weeks for 12 weeks. At Week 12, a secondary randomization occurred in Group 3 for those participants who completed the Week 12 assessments. After Week 12, dosing in Group 3 was monthly up to Week 28, then criteria based re-dosing from Week 28-52.
- Group 4: REGN2176-3 (3 mg:2 mg) to IAI 2 mg: Intravitreal injection of REGN2176-3 (REGN2176 3 mg and REGN3 2 mg) every 4 weeks for 12 weeks. At Week 12, a secondary randomization occurred in Group 2 for those participants who completed the Week 12 assessments. After Week 12, dosing in Group 4 was monthly with IAI 2 mg up to Week 28, then criteria based re-dosing from Week 28-52.
- Group 5: IAI 2 mg to REGN2176-3 (3 mg:2 mg): IAI every 4 weeks for 12 weeks. At Week 12, a secondary randomization occurred in Group 3 for those participants who completed the Week 12 assessments. After Week 12, dosing in Group 5 was monthly with REGN2176-3 (REGN2176 3 mg and REGN3 2 mg) up to Week 28, then criteria based re-dosing from Week 28-52.
Period: Period 1 (Day 1 to Week 12)
Arm/Group | Group 1: REGN2176-3 (1 mg:2 mg) | Group 2: REGN2176-3 (3 mg:2 mg) | Group 3: Intravitreal Aflibercept Injection (IAI) 2 mg | Group 4: REGN2176-3 (3 mg:2 mg) to IAI 2 mg | Group 5: IAI 2 mg to REGN2176-3 (3 mg:2 mg)
Started (Safety Analysis Set (SAF): all initially randomized participants who received any study drug) | 103; 103 Study Eyes | 200; 200 Study Eyes | 202; 202 Study Eyes | 0; 0 Study Eyes | 0; 0 Study Eyes
Completed (Completed week 12 in the SAF) | 101; 101 Study Eyes | 196; 196 Study Eyes | 200; 200 Study Eyes | 0; 0 Study Eyes | 0; 0 Study Eyes
Not Completed | 2; 2 Study Eyes | 4; 4 Study Eyes | 2; 2 Study Eyes | 0; 0 Study Eyes | 0; 0 Study Eyes
Not completed — Adverse Event | 0 | 2 | 0 | 0 | 0
Not completed — Death | 1 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0
Period: Period 2 (Day 1 to Week 52/End of Study)
Arm/Group | Group 1: REGN2176-3 (1 mg:2 mg) | Group 2: REGN2176-3 (3 mg:2 mg) | Group 3: Intravitreal Aflibercept Injection (IAI) 2 mg | Group 4: REGN2176-3 (3 mg:2 mg) to IAI 2 mg | Group 5: IAI 2 mg to REGN2176-3 (3 mg:2 mg)
Started (SAF (includes all initially randomized participants who received any study drug)) | 103; 103 Study Eyes | 106; 106 Study Eyes | 108; 108 Study Eyes | 94; 94 Study Eyes | 94; 94 Study Eyes
Completed (Completed week 52 in the SAF) | 70; 70 Study Eyes | 64; 64 Study Eyes | 71; 71 Study Eyes | 67; 67 Study Eyes | 67; 67 Study Eyes
Not Completed | 33; 33 Study Eyes | 42; 42 Study Eyes | 37; 37 Study Eyes | 27; 27 Study Eyes | 27; 27 Study Eyes
Not completed — Adverse Event | 3 | 7 | 6 | 2 | 2
Not completed — Death | 1 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 26 | 28 | 26 | 21 | 24
Not completed — Withdrawal by Subject | 3 | 4 | 4 | 1 | 0
Not completed — Lost to Follow-up | 0 | 2 | 1 | 2 | 1
Not completed — Other Un-specified | 0 | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline population included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: REGN2176-3 (1 mg:2 mg) | Group 2: REGN2176-3 (3 mg:2 mg) | Group 3: Intravitreal Aflibercept Injection (IAI) 2 mg | Total
Number analyzed (Participants) | 103 | 200 | 202 | 505
Age, Continuous [Mean (Standard Deviation); unit: years] | 79.2 (8.01) | 78.6 (8.77) | 77.7 (8.61) | 78.3 (8.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 121 | 135 | 317
  Male | 42 | 79 | 67 | 188
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 7 | 6 | 14
  Not Hispanic or Latino | 102 | 193 | 196 | 491
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 5 | 9 | 10 | 24
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 2 | 3
  White | 98 | 189 | 186 | 473
  More than one race | 0 | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 2 | 2
Region of Enrollment [Number; unit: Participants]
  United States | 98 | 193 | 194 | 485
  Japan | 5 | 7 | 8 | 20

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Best Corrected Visual Acuity (BCVA) of the Study Eye at Week 12
Description: Visual function of the study eye was assessed using the Early Treatment Diabetic Retinopathy Study (ETDRS) protocol at 4 meters. BCVA score was measured using an eye chart and was reported as the number of letters read correctly at a testing distance of 4 meters using the ETDRS Scale (ranging from 0 to 100 letters) in the study eye. The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). An increase in the number of letters read correctly means that vision has improved. Change from baseline calculated by subtracting baseline value from observed post-baseline value at Week 12.
Time Frame: Baseline, Week 12
Population: Full analysis set (FAS) that included all randomized participants who received any study treatment, had a baseline measurement of BCVA, and at least 1 post-baseline assessment of BCVA. Last observation carried forward (LOCF) method was used to impute missing data.
Measure: Least Squares Mean (Standard Error); unit: Letters
Arm/Group | Group 1: REGN2176-3 (1 mg:2 mg) | Group 2: REGN2176-3 (3 mg:2 mg) | Group 3: Intravitreal Aflibercept Injection (IAI) 2 mg
Number analyzed (Participants) | 103 | 200 | 202
Letters | 5.9 (1.01) | 5.7 (0.73) | 7.4 (0.72)
Statistical Analysis 1: Comparison: Group 1: REGN2176-3 (1 mg:2 mg) vs Group 3: Intravitreal Aflibercept Injection (IAI) 2 mg; To control for the family-wise type I error rate of 5%, for each of the 2 REGN2176-3 groups the 2-sided hypothesis comparing REGN2176-3 (1 mg: 2 mg) vs. Intravitreal Aflibercept Injection (IAI) 2 mg was tested at a significance level of α = 2.5%; Test type: Superiority — Analysis was performed using analysis of covariance (ANCOVA) model with baseline measurements as covariate and treatment group, baseline angiographic choroidal neovascularization (CNV) subtype (predominantly or minimally classic versus occult versus occult with no classic lesions) as fixed factors; p = 0.2052, ANCOVA — Threshold for significance at 0.025 level; Least Squares (LS) Mean Difference = -1.58, 95% CI 2-sided [-4.37 to 1.22]
Statistical Analysis 2: Comparison: Group 2: REGN2176-3 (3 mg:2 mg) vs Group 3: Intravitreal Aflibercept Injection (IAI) 2 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — Analysis was performed using ANCOVA model with baseline measurements as covariate and treatment group, baseline angiographic choroidal neovascularization (CNV) subtype (predominantly or minimally classic versus occult versus occult with no classic lesions) as fixed factors; p = 0.0982, ANCOVA — Threshold for significance at 0.025 level; Least Squares (LS) Mean Difference = -1.70, 95% CI 2-sided [-4.00 to 0.61]

2. Secondary Outcome: Change From Baseline in Central Subfield Retinal Thickness (CST) at Week 12, as Measured by Optical Coherence Tomography (OCT)
Description: CST was assessed using spectral domain optical coherence tomography (SD-OCT), a non-invasive diagnostic system providing high-resolution imaging sections of the retina. SD-OCT was performed in the study eye after pupil dilation. A negative change from baseline indicated improvement. Change from baseline calculated by subtracting baseline value from LOCF post-baseline value at Week 12.
Time Frame: Baseline, Week 12
Population: Analysis was performed on FAS. LOCF method was used to impute missing data.
Measure: Least Squares Mean (Standard Error); unit: Microns
Arm/Group | Group 1: REGN2176-3 (1 mg:2 mg) | Group 2: REGN2176-3 (3 mg:2 mg) | Group 3: Intravitreal Aflibercept Injection (IAI) 2 mg
Number analyzed (Participants) | 103 | 200 | 202
Microns | -131.1 (6.88) | -116.9 (4.96) | -134.4 (4.92)

3. Secondary Outcome: Percentage of Participants With Complete Resolution of Intraretinal and Subretinal Fluid From Baseline at Week 12 Measured by Optical Coherence Tomography (OCT)
Description: CST was assessed using spectral domain optical coherence tomography (SD-OCT), a non-invasive diagnostic system providing high-resolution imaging sections of the retina. SD-OCT was performed in the study eye after pupil dilation.
Time Frame: Week 12
Population: Analysis was performed on FAS. LOCF method was used to impute missing data.
Measure: Number; unit: Percentage of Participants
Arm/Group | Group 1: REGN2176-3 (1 mg:2 mg) | Group 2: REGN2176-3 (3 mg:2 mg) | Group 3: Intravitreal Aflibercept Injection (IAI) 2 mg
Number analyzed (Participants) | 103 | 200 | 202
Percentage of Participants | 35.0 | 24.0 | 42.1

4. Secondary Outcome: Change From Baseline in Choroidal Neovascularization (CNV) Area at Week 12 Measured by Fluorescein Angiography (FA)
Description: The anatomical state of the retinal vasculature of the study eye and the fellow eye was evaluated by funduscopic examination, fundus photography and FA to evaluate the total lesion area, CNV area, classic CNV area, and fluorescein leakage. CNV area values measured in square millimeters, each disc area was equivalent to 2.54 mm^2 on the retina; lower values represent better outcomes.
Time Frame: Baseline, Week 12
Population: Analysis was performed on FAS. LOCF was used to impute missing data. Here, number of participants analyzed = participants with available data for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Square Millimeter (mm^2)
Arm/Group | Group 1: REGN2176-3 (1 mg:2 mg) | Group 2: REGN2176-3 (3 mg:2 mg) | Group 3: Intravitreal Aflibercept Injection (IAI) 2 mg
Number analyzed (Participants) | 97 | 187 | 192
Square Millimeter (mm^2) | -3.4 (0.44) | -2.0 (0.31) | -3.6 (0.31)

5. Secondary Outcome: Change From Baseline in Total Lesion Size at Week 12 Measured by Fluorescein Angiography (FA)
Description: Total Lesion Size was assessed by Fluorescein Angiography.
Time Frame: Baseline, Week 12
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Group 1: REGN2176-3 (1 mg:2 mg) | Group 2: REGN2176-3 (3 mg:2 mg) | Group 3: Intravitreal Aflibercept Injection (IAI) 2 mg
Number analyzed (Participants) | 97 | 187 | 192
mm | -3.1 (0.43) | -2.1 (0.31) | -3.5 (0.31)

6. Secondary Outcome: Percentage of Participants Who Gained At Least 15 Letters in BCVA From Baseline at Week 12, Measured by 4-meter Early Treatment Diabetic Retinopathy Scale (ETDRS)
Description: Visual function of the study eye was assessed using the Early Treatment Diabetic Retinopathy Study (ETDRS) protocol at 4 meters. BCVA score was measured using an eye chart and was reported as the number of letters read correctly at a testing distance of 4 meters using the ETDRS Scale (ranging from 0 to 100 letters) in the study eye. The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). An increase in the number of letters read correctly means that vision has improved. This outcome assessed the percentage of participants who gained 15 or more letters of visual acuity at Week 12 compared with baseline.
Time Frame: Week 12
Population: Analysis was performed on FAS. LOCF was used to impute missing data.
Measure: Number; unit: Percentage of Participants
Arm/Group | Group 1: REGN2176-3 (1 mg:2 mg) | Group 2: REGN2176-3 (3 mg:2 mg) | Group 3: Intravitreal Aflibercept Injection (IAI) 2 mg
Number analyzed (Participants) | 103 | 200 | 202
Percentage of Participants | 11.7 | 18.5 | 21.8

7. Secondary Outcome: Percent Change From Baseline in Subretinal Hyperreflectivity Material (SHM) at Week 12 Measured by Optical Coherence Tomography (OCT)
Description: SHM was assessed using spectral domain optical coherence tomography (SD-OCT), a non-invasive diagnostic system providing high-resolution imaging sections of the retina. SD-OCT was performed in the study eye after pupil dilation. A negative change from baseline indicated improvement.
Time Frame: Baseline, Week 12
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Group 1: REGN2176-3 (1 mg:2 mg) | Group 2: REGN2176-3 (3 mg:2 mg) | Group 3: Intravitreal Aflibercept Injection (IAI) 2 mg
Number analyzed (Participants) | 94 | 191 | 193
Percent change | -50.0 (5.94) | -41.9 (4.17) | -48.8 (4.14)

8. Secondary Outcome: Change From Baseline in Central Retinal/Lesion Thickness at Week 12 Measured by Optical Coherence Tomography (OCT)
Description: as for outcome 2
Time Frame: Baseline, Week 12
Population: Analysis was performed on FAS. LOCF was used to impute missing data.
Measure: Least Squares Mean (Standard Error); unit: Microns
Arm/Group | Group 1: REGN2176-3 (1 mg:2 mg) | Group 2: REGN2176-3 (3 mg:2 mg) | Group 3: Intravitreal Aflibercept Injection (IAI) 2 mg
Number analyzed (Participants) | 103 | 200 | 202
Microns | -150.7 (7.40) | -139.6 (5.32) | -160.4 (5.29)

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) were collected from signature of the informed consent form up to the final visit (Week 52) regardless of seriousness or relationship to investigational product.
Description: Reported AEs are treatment-emergent and are defined as AEs starting after the first study eye injection and no later than 30 days after the last study eye or fellow eye injection. Analysis was performed on safety analysis set (SAF) and included all initially randomized participants who received any study drug before Week 12; it was based on Week 12 secondary randomization group assignment.
Arm/Group | Group 1: REGN2176-3 (1 mg:2 mg) | Group 2: REGN2176-3 (3 mg:2 mg) | Group 3: Intravitreal Aflibercept Injection (IAI) 2 mg | Group 4: REGN2176-3 (3 mg:2 mg) to IAI 2 mg | Group 5: IAI 2 mg to REGN2176-3 (3 mg:2 mg)
All-Cause Mortality (participants affected / at risk) | 3/103 | 2/106 | 3/108 | 1/94 | 1/94
Serious Adverse Events (participants affected / at risk) | 17/103 | 20/106 | 23/108 | 17/94 | 15/94
Other Adverse Events (participants affected / at risk) | 48/103 | 50/106 | 51/108 | 52/94 | 52/94
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: REGN2176-3 (1 mg:2 mg) (N=103) | Group 2: REGN2176-3 (3 mg:2 mg) (N=106) | Group 3: Intravitreal Aflibercept Injection (IAI) 2 mg (N=108) | Group 4: REGN2176-3 (3 mg:2 mg) to IAI 2 mg (N=94) | Group 5: IAI 2 mg to REGN2176-3 (3 mg:2 mg) (N=94)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 4 (4) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardio-Respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ischaemic cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stress cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blindness (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Study eye
Blindness transient (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Study eye
Macular degeneration (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Study eye
Neovascular age-related macular degeneration (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Study eye
Open angle glaucoma (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Study eye
Retinal haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) — Study eye
Uveitis (Eye disorders) | 1 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) — Study eye
Visual acuity reduced (Eye disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) — Study eye
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-Cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Endophthalmitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Study eye
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infectious colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Vestibular neuronitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Comminuted fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Impacted fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lip squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Non-Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prostate cancer stage ii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Study eye
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Basal ganglia stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dementia alzheimer's type (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Major depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Calculus ureteric (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neovascular age-related macular degeneration (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Fellow eye
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: REGN2176-3 (1 mg:2 mg) (N=103) | Group 2: REGN2176-3 (3 mg:2 mg) (N=106) | Group 3: Intravitreal Aflibercept Injection (IAI) 2 mg (N=108) | Group 4: REGN2176-3 (3 mg:2 mg) to IAI 2 mg (N=94) | Group 5: IAI 2 mg to REGN2176-3 (3 mg:2 mg) (N=94)
Cataract (Eye disorders) | 6 (6) | 1 (1) | 2 (2) | 1 (1) | 0 (0) — Fellow eye
Conjunctival haemorrhage (Eye disorders) | 6 (6) | 4 (4) | 6 (7) | 11 (13) | 9 (12) — Study eye
Eye pain (Eye disorders) | 3 (3) | 5 (6) | 1 (1) | 6 (9) | 2 (2) — Study eye
Neovascular age-related macular degeneration (Eye disorders) | 1 (1) | 10 (10) | 8 (9) | 8 (8) | 5 (5) — Fellow eye
Posterior capsule opacification (Eye disorders) | 1 (1) | 2 (2) | 1 (1) | 4 (4) | 5 (5) — Study eye
Retinal haemorrhage (Eye disorders) | 6 (7) | 8 (8) | 3 (3) | 5 (5) | 3 (3) — Study eye
Vitreous detachment (Eye disorders) | 3 (3) | 3 (4) | 2 (2) | 7 (7) | 3 (3) — Study eye
Vitreous floaters (Eye disorders) | 2 (3) | 1 (1) | 1 (1) | 3 (3) | 10 (15) — Study eye
Nasopharyngitis (Infections and infestations) | 3 (3) | 6 (6) | 9 (12) | 5 (5) | 8 (8)
Sinusitis (Infections and infestations) | 2 (3) | 7 (8) | 2 (2) | 4 (4) | 7 (7)
Urinary tract infection (Infections and infestations) | 7 (8) | 7 (9) | 4 (4) | 7 (8) | 13 (17)
Fall (Injury, poisoning and procedural complications) | 5 (6) | 6 (6) | 2 (2) | 4 (4) | 3 (3)
Hypertension (Vascular disorders) | 6 (6) | 4 (4) | 10 (10) | 2 (2) | 5 (6)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0) | 2 (2) | 2 (2) | 6 (7)
Posterior capsule opacification (Eye disorders) | 5 (5) | 1 (1) | 2 (2) | 5 (5) | 2 (3) — Fellow eye
Vitreous floaters (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 4 (5) | 5 (5) — Fellow eye

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator has the right to independently publish study results from the investigator's site after a multi-center publication, or a defined period after the completion of the study by all sites. The investigator must provide the sponsor a copy of any such publication derived from the study for review and comment in advance of any submission, and delay publication, if requested, to allow the Sponsor to preserve its proprietary rights.